CLINICAL TRIAL: NCT04061278
Title: A Multicenter, Prospective, Phase III Randomized Controlled Clinical Study Comparing 4 Cycles of Neoadjuvant Chemotherapy Combined With Radiotherapy Versus 3cycles of Neoadjuvant Chemotherapy Combined With Concurrent Chemoradiotherapy for the Treatment of N2-3 Nasopharyngeal Carcinoma
Brief Title: A Multicenter, Prospective, Phase III Randomized Controlled Clinical Study for the Treatment of N2-3 Nasopharyngeal Carcinoma Patients
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Second Affiliated Hospital, School of Medicine, Zhejiang University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: SAHZhejiangU-2019-009
Record Dates: First submitted 2019-08-13; First posted 2019-08-19 (Actual); Last update posted 2020-05-12 (Actual); Status verified 2019-08

CONDITIONS: Nasopharyngeal Carcinoma; Neoadjuvant Chemotherapy
Keywords: Nasopharyngeal Carcinoma; Neoadjuvant Chemotherapy; Concurrent Chemoradiotherapy
MeSH Terms: conditions — Nasopharyngeal Carcinoma | interventions — Chemoradiotherapy

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- 4 Cycles of Neoadjuvant Chemotherapy With Radiotherapy (Experimental): Four cycles of neoadjuvant chemotherapy combined with radical radiotherapy
  Interventions: Drug: 4 cycles of Neoadjuvant Chemotherapy With Definitive Radiotherapy
- 3cycles of Neoadjuvant Chemotherapy With chemoradiotherapy (Active Comparator): 3 cycles of Neoadjuvant Chemotherapy Combined With Concurrent Chemoradiotherapy
  Interventions: Drug: 3 cycles of Neoadjuvant Chemotherapy With concurrent chemoradiotherapy

INTERVENTIONS:
Drug: 4 cycles of Neoadjuvant Chemotherapy With Definitive Radiotherapy — 4 Cycles of Neoadjuvant Chemotherapy With Definitive Radiotherapy, instead of Concurrent Chemoradiotherapy
  Arms: 4 Cycles of Neoadjuvant Chemotherapy With Radiotherapy
Drug: 3 cycles of Neoadjuvant Chemotherapy With concurrent chemoradiotherapy — 3 cycles of Neoadjuvant Chemotherapy With concurrent chemoradiotherapy, instead of definitive radiotherapy
  Arms: 3cycles of Neoadjuvant Chemotherapy With chemoradiotherapy

SUMMARY:
At the initial diagnosis of locally advanced nasopharyngeal carcinoma, a considerable proportion of patients have developed distant metastasis, forming subclinical lesions. Nowadays, with the advent of intensity modulated radiotherapy, the local-regional area is under well controlled. However, distant metastasis is still the main cause of failure in treatment of stage N2-3 nasopharyngeal carcinoma.The severe toxicity of synchronous chemotherapy and the dose intensity of single drug is not enough to effectively control existing subclinical lesions. Neoadjuvant chemotherapy with sufficient intensity (four cycles) can possible effectively kill subclinical lesions prior to the initiation of concurrent chemoradiotherapy, thereby reducing distant metastasis of stage N2-3 nasopharyngeal carcinoma. Meanwhile, four cycles of chemotherapy have been shown to be well tolerated in other tumors. In conclusion, 4-cycle neoadjuvant chemotherapy in combination with radiotherapy is expected to further control the distant metastasis rate of N2-3 nasopharyngeal carcinoma and improve the survival rate.

ELIGIBILITY:
Inclusion Criteria:

1. Non-keratinizing nasopharyngeal carcinoma diagnosed by pathology;
2. According to the UICC/AJCC eighth edition staging criteria, clinical staging was T1-4N2 -3M0 (stage N2-3 nasopharyngeal carcinoma);
3. Patients who have not received disease-related anti-tumor system therapy;
4. Age 18~70 years;
5. Perfect liver and kidney function: total bilirubin ≤1.5 times the upper limit of normal value (ULN); AST and ALT≤2.5 ULN; Alkaline phosphatase ≤2.5 ULN; Creatinine clearance rate ≥80 mL/min;
6. Complete blood system function: neutrophil count (ANC) ≥2×109/L, platelet count ≥100×109/L and hemoglobin ≥9 g/dL;
7. Cartesian score ≥70; or ECOG PS 0 or 1
8. Prior to enrollment, the patients must undergo nasopharynx + neck MRI, chest + upper abdomen CT, ECT and other examinations of the whole body bone.
9. Sign the informed consent.

Exclusion Criteria:

1. Patients with distant metastases were identified at the time of diagnosis;
2. Patients with severe medical complications, severe organ (heart, lung) dysfunction, or neuropsychiatric disorders at the time of diagnosis;
3. Previous cases of other malignancies;Complicated with other malignant tumors;Except for cured basal cell carcinoma of the skin or squamous cell carcinoma of the skin or carcinoma in situ of any other site;
4. Use any other investigational drug or participate in another clinical trial with therapeutic intent within 3 months prior to enrollment;
5. A woman who is pregnant or lactating;
6. Known active HIV or HBV, HCV infection;
7. Known to be allergic to drugs that may be used;
8. The researchers did not consider participants to be eligible for this study.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 246 (Estimated)
Dates: Start 2019-08-01 (Actual); Primary Completion 2022-06-30 (Estimated); Study Completion 2022-12-31 (Estimated)

PRIMARY OUTCOMES:
5-year overall survival | 5 years
  the duration between the date of diagnosed and date of patient death
5-year metastatic free survival | 5 years
  the duration between the date of diagnosed and date of metastasis

SECONDARY OUTCOMES:
5-year disease-free survival | 5 years
  the duration between the date of diagnosed and date of related disease
5-year recurrence-free survival | 5 years
  the duration between the date of diagnosed and date of recurrence
Safety (incidence of grade 3/4 adverse reactions) | 5 years
  treatment related toxic effects

CONTACTS AND LOCATIONS:
Overall Officials: Qichun Wei, Study Chair — 2nd Affiliated Hospital, School of Medicine, Zhejiang University, China
Locations (12):
- China (12):
  - Fujian Medical University Union Hospital, Fuzhou, Fujian
  - Cancer prevention and treatment center, sun yat-sen university, Guandong, Guangdong
  - The first affiliated hospital, college of medicinle, Zhejiang University, Hangzhou, Zhejiang
  - Zhejiang Cancer Hospital, Hangzhou, Zhejiang
  - Zhejiang Provincial People's Hospital, Hangzhou, Zhejiang
  - 2nd Affiliated Hospital, School of Medicine, Zhejiang University, China, Hangzhou, Zhejiang
  - Zhejiang Xiaoshan Hospital, Hangzhou, Zhejiang
  - Jinhua Central Hospital, Jinhua, Zhejiang
  - Lishui City Central Hospital, Lishui, Zhejiang
  - Ningbo Yinzhou People's Hospital, Ningbo, Zhejiang
  - Ningbo No.2 Hospital, Ningbo, Zhejiang
  - People's Hospital of Quzhou, Quzhou, Zhejiang